CLINICAL TRIAL: NCT03092310
Title: Feasibility Evaluation of an Artificial Pancreas With an Enhanced Model Predictive Control (eMPC) Controller and a Health Monitoring System (HMS) With a Glucose Prediction Trust Index
Brief Title: Feasibility Evaluation of an Artificial Pancreas With Glucose Prediction Trust Index
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sansum Diabetes Research Institute (Other)
Collaborators: Harvard University (Other)
Responsible Party: Principal Investigator, Jordan Pinsker, Research Physician, Sansum Diabetes Research Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00020556
Record Dates: First submitted 2017-03-15; First posted 2017-03-27 (Actual); Last update posted 2018-07-12 (Actual); Status verified 2018-07

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Artificial Pancreas
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Pancreas, Artificial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Artificial Pancreas (Experimental): The artificial pancreas device will employ its enhanced Model Predictive Control (MPC) algorithm with a target glucose level of 110 mg/dL with a trust index for MPC-predicted glucose values, weighing future glucose predictions and only acting on predictions with higher weight in the trust index. The Health Monitoring System algorithm uses the same CGM data as the MPC control algorithm but utilizes a separate algorithm for trending and predictions of future glucose values. Using a redundant and independent algorithm is an important safety feature of the overall AP device.
  Interventions: Device: Artificial Pancreas Device

INTERVENTIONS:
Device: Artificial Pancreas Device — Artificial Pancreas Device

SUMMARY:
The purpose of this pilot study is to establish that closed-loop insulin delivery with a target enchanted model predictive control (eMPC)/Health Monitoring System (HMS) algorithms with a trust index of the predicted glucose value is safe and effective, to analyze and learn to improve upon the accuracy of the predicted glucose values, and to collect efficacy data to inform a future larger study.

DETAILED DESCRIPTION:
This is a feasibility study of an artificial pancreas (AP) system with our previously validated target eMPC and HMS algorithms, with the addition of a trust index of the predicted glucose value integrated into the portable Artificial Pancreas System (pAPS). The system will be evaluated on up to 20 subjects, with the goal of 10 subjects completing a 48-hour closed-loop session at one clinical site (William Sansum Diabetes Center). During the session subjects will bolus for all meals and snacks and perform a 45-minute walking session.

The purpose of this pilot study is to establish that closed-loop insulin delivery with a target enchanted model predictive control (eMPC)/Health Monitoring System (HMS) algorithms with a trust index of the predicted glucose value is safe and effective, to analyze and learn to improve upon the accuracy of the predicted glucose values, and to collect efficacy data to inform a future larger study.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 and ≤ 75 years at the time of screening.
* Clinical diagnosis of type 1 diabetes for at least one year.
* Has been using an insulin pump for at least 6 months at the time of screening.
* HbA1c < 10%, as performed by point of care or central laboratory testing. A1c will be assessed at the screening visit, or if already completed within 2 months of the screening visit, the prior lab value may be used in lieu of repeating this assessment.
* Serum creatinine of < 2.0 mg/dL. Serum creatinine will be assessed at the screening visit, or if already completed within 2 months of the screening visit, the prior lab value may be used in lieu of repeating this assessment.
* Bolus for all meals and snacks that contain ≥ 5 grams of carbohydrate.
* Willing to perform at least 7 fingerstick blood glucose tests a day.
* Willing to refrain from taking acetaminophen products for the duration of the clinical trial. If acetaminophen is taken, subject is to avoid making any insulin dosing decisions based on CGM for at least 12 hours.
* Willing to abide by the study protocol and use study-provided devices, including the Omnipod, Dexcom CGM, glucometer, ketone meter and pAPS tablet.

Exclusion Criteria:

* Pregnancy
* One or more episodes of hypoglycemia requiring an emergency room visit or hospitalization in the past 6 months.
* One or more episodes of hyperglycemia requiring an emergency room visit or hospitalization in the past 6 months.
* Known unstable cardiac disease or untreated cardiac disease, as revealed by history or physical examination.
* Dermatological conditions that would preclude wearing a CGM sensor or Pod.
* One or more seizures in the past year.
* Screening A1c ≥ 10% or serum creatinine ≥ 2.0 mg/dL.
* Any condition that could interfere with participating in the trial, based on investigator judgment.
* Concurrent use of any non-insulin glucose-lowering agent (including GLP-1 agonists, Symlin, DPP-4 inhibitors, SGLT-2 inhibitors, biguanides, sulfonylureas and naturaceuticals), defined as using any of these medications within 30 days of the screening visit or during the study.
* Participation in another pharmaceutical or device trial at the time of enrollment or during the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-03-20 (Actual); Primary Completion 2017-12-20 (Actual); Study Completion 2017-12-20 (Actual)

PRIMARY OUTCOMES:
Percent time within the target glucose range of 70-180 mg/dl overall as assessed by continuous glucose monitoring (CGM). | 48 hours
  The primary endpoint for this pilot study will be time within the target glucose range of 70-180 mg/dl overall as assessed by continuous glucose monitoring (CGM), during closed-loop use, determining if the combination of eMPC and the assessment of trust index can provide safe and effective glucose control.

SECONDARY OUTCOMES:
Assessment of the trust index predictions vs. standard eMPC glucose predictions. | 48 hours
  During closed-loop use, assessment of the trust index predictions vs. standard eMPC glucose predictions (frequency of moving away from nominal weights of predicted glucose).
Frequency of hypoglycemia during closed-loop use. | 48 hours
  Frequency of hypoglycemia during closed-loop use, defined as percent time glucose is below predefined thresholds of 70 mg/dl, 60 mg/dl and 50 mg/dL.
Frequency of hyperglycemia during closed-loop use. | 48 hours
  Frequency of hyperglycemia during closed-loop use, defined as percent time glucose is above predefined thresholds of 180 mg/dl, 250 mg/dl, and 300 mg/dL.
Percent time within the target glucose range of 70-140 mg/dl during closed-loop use. | 48 hours
  Percent time within the target glucose range of 70-140 mg/dl overall as assessed by continuous glucose monitoring (CGM), during closed-loop use.
Percent time glucose is within range 70-150 mg/dl postprandial within 5 hours following meals, during closed-loop use. | 48 hours
  Percent time glucose is within range 70-150 mg/dl postprandial within 5 hours following meals, during closed-loop use.
Standard Deviation and Coefficient of Variation of glucose values | 48 hours
  To measure glycemic variability, the standard deviation and coefficient of variation of glucose values (as measured by continuous glucose monitoring) will be determined during the 48 hours of closed-loop use.
Markers of hypo- and hyperglycemia | 48 hours
  Markers of hypo- and hyperglycemia, to include LBGI (Low blood glucose index) and HBGI (High blood glucose index), during closed-loop use.
Insulin Doses Given | 48 hours
  Change in total daily doses and post prandial insulin doses given during the 48 hours of closed-loop use.
Number of treatments given for hypoglycemia (defined as carbohydrates given for treatment of a documented or suspected low blood sugar), during the 48 hours of closed-loop use. | 48 hours
  Treatments for hypoglycemia given during the 48 hours of closed-loop use. Hypoglycemia treatments may be given in response to alerts from the HMS, if blood glucose < 70 mg/dL, or at the request of the subject or investigator.
Number of alerts given by the HMS to prevent hypoglycemia | 48 hours
  Number of alerts given by the HMS to prevent hypoglycemia during closed-loop use.
Failure analysis of the devices/connectivity issues that may occur (# disconnects and device restarts). | 48 hours
  Failure analysis of the devices/connectivity issues that may occur during closed-loop use. This includes number of CGM communication losses with 3 or more missed points, and number of times the entire system required a restart.

CONTACTS AND LOCATIONS:
Overall Officials: Jordan E Pinsker, MD, Principal Investigator — Sansum Diabetes Research Institute; Eyal Dassau, PhD, Principal Investigator — Harvard John A. Paulson School of Engineering and Applied Sciences, Harvard University; Francis J Doyle III, PhD, Principal Investigator — Harvard John A. Paulson School of Engineering and Applied Sciences, Harvard University; Alejandro Leguna, PhD, Principal Investigator — Harvard John A. Paulson School of Engineering and Applied Sciences, Harvard University
Locations (1):
- William Sansum Diabetes Center, Santa Barbara, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Pinsker JE, Laguna Sanz AJ, Lee JB, Church MM, Andre C, Lindsey LE, Doyle FJ 3rd, Dassau E. Evaluation of an Artificial Pancreas with Enhanced Model Predictive Control and a Glucose Prediction Trust Index with Unannounced Exercise. Diabetes Technol Ther. 2018 Jul;20(7):455-464. doi: 10.1089/dia.2018.0031. PMID 29958023